CLINICAL TRIAL: NCT02219360
Title: Treatment in Patients Hospitalized With Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Acronym: TripAE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Wang Ying, resident, Beijing Chao Yang Hospital
Other Study IDs: 2014-K-115
Record Dates: First submitted 2014-07-09; First posted 2014-08-18 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: acute; exacerbation; chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 25-(OH)-VD3 and glycated albumin will be tested
Oversight: Data Monitoring Committee: No

SUMMARY:
Chronic obstructive pulmonary disease has become a serious global health care and public health problems due to its high prevalence, high morbidity and heavy economic burden. Acute exacerbation of chronic obstructive pulmonary disease is one of the most important causes of death in patients with COPD. Systemic corticosteroids therapy is recommended in COPD exacerbations. In clinical practice for the treatment of acute exacerbation of COPD， antibiotic application is still controversial. Evidence from current guideline is based on strict criteria from randomized controlled trials, thus the given condition is simplified. Patients meet the criteria account for the minority in the real world. Therefore, it is still not clear whether most patients benefit from the recommended treatment. In our design, hospitalized patients with acute exacerbation of COPD will be enrolled, with their treatment, arterial hypoxemia, recovery time and length of hospitalization being observed. The main purpose is to evaluate the benefit effect of current recommended treatment of acute exacerbation of COPD in the real world.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease has become a serious global health care and public health problems due to its high prevalence, high morbidity and heavy economic burden. Acute exacerbation of COPD is one of the most important causes of death in patients with COPD. The global strategy for the diagnosis, management, and prevention of COPD recommends systemic corticosteroids therapy in COPD exacerbations as it can shorten recovery time, reduce treatment failure, improve lung function and arterial hypoxemia. In clinical practice for the treatment of acute exacerbation of COPD， antibiotic application is still controversial. Evidence from current guideline is based on strict criteria from randomized controlled trials, thus the given condition is simplified. Patients meet the criteria account for the minority in the real world. Therefore, it is still not clear whether most patients benefit from the recommended treatment. In our design, hospitalized patients with acute exacerbation of COPD will be enrolled, with their treatment, arterial hypoxemia, recovery time and length of hospitalization being observed. The main purpose is to evaluate the benefit effect of current recommended treatment of acute exacerbation of COPD in the real world.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with acute exacerbation of chronic obstructive pulmonary disease
* Age≥ 40years old

Exclusion Criteria:

* The first diagnosis which caused hospitalization is not acute exacerbation of chronic obstructive pulmonary disease
* Chest radiography shows congestive heart failure
* Chest CT shows lung cancer, active pulmonary tuberculosis, pulmonary thromboembolism or interstitial lung diseases
* Serious cardiac failure, renal insufficiency or hepatic dysfunction

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized with acute exacerbation of chronic obstructive pulmonary disease from 1st July, 2014 from Beijing Chao Yang Hospital
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-06 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
change of the score of COPD Assesment Test as a measurement of the overall condition of the patient | baseline, 1 month after dischahge, 2 months after discharge

SECONDARY OUTCOMES:
change of the score of modified Medical British Research Council questionaire as a measurement of the overall condition of the patient | baseline, 1 month after discharge, 2 months after discharge

OTHER OUTCOMES:
percentage of use of systemic corticosteroid in patients | 8 months after the first enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Wang Ying, Master, Principal Investigator — Beijing Chao Yang Hospital; Huang Kewu, M.D., Study Chair — Beijing Chao Yang Hospital